CLINICAL TRIAL: NCT04731467
Title: A Phase 1/2 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of CM24 in Combination with Nivolumab in Adults with Advanced Solid Tumors
Brief Title: A Study of CM24 in Combination with Nivolumab in Adults with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Famewave Ltd. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Purple Biotech Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FW-2020-1
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer; Pancreatic Cancer; Ovarian Cancer; Papillary Thyroid Cancer; Melanoma; Colorectal Adenocarcinoma
Keywords: CM24; nivolumab; Opdivo; nab-paclitaxel; Abraxane
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Ovarian Neoplasms; Thyroid Cancer, Papillary; Melanoma | interventions — Nivolumab; Taxes

STUDY DESIGN:
Masking Description: Parts A and C are non-randomized parts, part D is a randomized part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A- Dose escalation of CM24 in combination with nivolumab (Experimental)
  Interventions: Drug: CM-24 and Nivolumab - Dose Escalation
- Part C- Expansion cohort of CM24 in combination with nivolumab, nab-paclitaxel and gemcitabine (Experimental)
  Interventions: Drug: CM-24, Nivolumab, Nab paclitaxel and Gemcitabine - Expansion
- Part C- Expansion cohort of CM24 in combination with nivolumab and Nal-IRI/5-FU/LV (Experimental)
  Interventions: Drug: CM-24, Nivolumab, and Nal-IRI/5-FU/LV - Expansion
- Part D- Expansion cohort of CM24 in combination with nivolumab, nab-paclitaxel and gemcitabine (Experimental)
  Interventions: Drug: CM-24, Nivolumab, Nab paclitaxel and Gemcitabine - Expansion
- Part D- Expansion cohort of CM24 in combination with nivolumab and Nal-IRI/5-FU/LV (Experimental)
  Interventions: Drug: CM-24, Nivolumab, and Nal-IRI/5-FU/LV - Expansion
- Part D- Expansion cohort of nivolumab in combination with nab-paclitaxel and gemcitabine (Active Comparator)
  Interventions: Drug: Nivolumab, Nab paclitaxel and Gemcitabine - Expansion
- Part D- Expansion cohort of nivolumab in combination with Nal-IRI/5-FU/LV (Active Comparator)
  Interventions: Drug: Nivolumab and Nal-IRI/5-FU/LV - Expansion

INTERVENTIONS:
Drug: CM-24 and Nivolumab - Dose Escalation — Dose escalation of CM24 with nivolumab in adult patients with selected recurrent or metastatic solid tumors
  Arms: Part A- Dose escalation of CM24 in combination with nivolumab
Drug: CM-24, Nivolumab, Nab paclitaxel and Gemcitabine - Expansion — Expansion cohort of CM24 in combination with nivolumab, nab-paclitaxel and gemcitabine in adult patients with advanced metastatic pancreatic cancer
  Arms: Part C- Expansion cohort of CM24 in combination with nivolumab, nab-paclitaxel and gemcitabine; Part D- Expansion cohort of CM24 in combination with nivolumab, nab-paclitaxel and gemcitabine
Drug: CM-24, Nivolumab, and Nal-IRI/5-FU/LV - Expansion — Expansion cohort of CM24 in combination with nivolumab and Nal-IRI/5-FU/LV in adult patients with advanced metastatic pancreatic cancer
  Arms: Part C- Expansion cohort of CM24 in combination with nivolumab and Nal-IRI/5-FU/LV; Part D- Expansion cohort of CM24 in combination with nivolumab and Nal-IRI/5-FU/LV
Drug: Nivolumab, Nab paclitaxel and Gemcitabine - Expansion — Expansion cohort of nivolumab in combination with nab-paclitaxel and gemcitabine in adult patients with advanced metastatic pancreatic cancer
  Arms: Part D- Expansion cohort of nivolumab in combination with nab-paclitaxel and gemcitabine
Drug: Nivolumab and Nal-IRI/5-FU/LV - Expansion — Expansion cohort of nivolumab in combination with Nal-IRI/5-FU/LV in adult patients with advanced metastatic pancreatic cancer
  Arms: Part D- Expansion cohort of nivolumab in combination with Nal-IRI/5-FU/LV

SUMMARY:
This is an open-label, multicenter, multi-dose escalation and dose expansion study in subjects with selected advanced solid tumors (Part A) and advanced metastatic pancreatic cancer (Parts C & D) to evaluate the safety and tolerability of CM-24 in combination with nivolumab. In Part C of the study gemcitabine/nab-paclitaxel or Nal-IRI/5-FU/LV will be administered subsequent to CM24 and nivolumab. CM24, nivolumab and gemcitabine/nab-paclitaxel or Nal-IRI/5-FU/LV are administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Previously treated subjects with recurrent and/or metastatic NSCLC, pancreatic cancer, ovarian cancer, papillary thyroid cancer, colorectal adenocarcinoma and melanoma with documented progression/intolerance following at least one previous therapy (and not more than 2 previous regimens); Part C: Subjects with histologically confirmed advanced metastatic pancreatic adenocarcinoma as defined by NCCN Guidelines; Subjects with islet cell neoplasms are excluded; subjects with a maximum of 1 prior treatment regimen for metastatic disease excluding: nab-paclitaxel containing regimens and up to 8 weeks from last chemotherapy treatment (Arm #1); fluoropyrimidine or irinotecan containing regimens and up to 8 weeks from last chemotherapy treatment (Arm #2).

   Part C, D: Subjects with histologically confirmed advanced metastatic pancreatic adenocarcinoma as defined by NCCN Guidelines; Subjects with islet cell neoplasms are excluded.
2. Parts C, D: Subjects who have progressed on or after standard of care chemotherapy with a maximum of 1 prior treatment regimen for advanced metastatic disease:

   * Subjects enrolled in arm with gemcitabine/nab-paclitaxel combination should have received a fluoropyrimidine and/or irinotecan containing regimen in the first line of treatment; Prior gemcitabine containing regimen may be allowed only if completed at least 6 months prior to study enrollment.
   * Arm #2: Subjects enrolled in arm with Nal-IRI/5FU/LV combination should have received a gemcitabine and/or nab-paclitaxel containing regimen in the first line of treatment; Prior irinotecan and/or fluoropyrimidine containing regimens may be allowed only if completed at least 6 months prior to study enrollment.
3. Part A: Availability of an archival tumor sample prior to first treatment. Parts C, D: Fresh tumor biopsy must be obtained within 3 months prior to enrollment and after the last systemic treatment was completed.
4. Must have at least 1 measurable lesion per RECIST1.1 with progressing or new tumors since last antitumor therapy;
5. ECOG performance status score of 0 or 1;
6. Adequate safety lab results;
7. Stable brain metastases;
8. WCBP (Women of Childbearing Potential) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test, WCBP must agree to abstain from sex or use an adequate method of contraception, males must abstain from sex with WCBP or use an adequate method of contraception.

Exclusion Criteria:

1. Part A: Received more than two prior systemic regimens for the metastatic disease Parts C and D: Received more than 1 prior systemic regimens for the advanced metastatic disease
2. Part A: History of weight loss >10% over the 2 months prior to Screening;
3. Unresolved AEs > Grade 1 from prior anticancer therapy.
4. Concurrent malignancy requiring treatment;
5. Active, untreated central nervous system (CNS) metastases;
6. Subjects previously treated with an anti PD-1/PD-L1 targeting agent with history immune mediated toxicity;
7. Severely immunocompromised;
8. History of allergy or hypersensitivity to any of the study treatment components;
9. Major surgery within 4 weeks of study administration;
10. Received a live / attenuated vaccine within 30 days of first treatment
11. Clinically relevant serious co-morbid medical conditions including, but not limited to:

    * Active infection;
    * Recent (within six months of Screening) cardiac disease, myocardial infarction, or severe or unstable angina;
    * History of serious arrhythmia;
    * Chronic obstructive or chronic restrictive pulmonary disease, pulmonary hypertension history of or active interstitial lung disease or pneumonitis;
    * Prior organ allograft;
    * Subjects with active, known or suspected autoimmune disease;
    * History of active or latent tuberculosis infection;
    * Positive test for HIV, HBV, or HCV;
12. Radiation within two weeks prior to the first study treatment;
13. Treatment with another investigational therapy within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer;
14. Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to treatment;
15. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of treatment emergent adverse events | Up to 24 months
  Incidence of treatment emergent adverse events with CM-24 and nivolumab in adults with selected recurrent or metastatic solid tumors
Part C: Safety and tolerability | Up to 24 months
  Incidence of treatment emergent adverse events with CM-24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV in adults with advanced metastatic pancreatic cancer
Part D: Overall survival | Up to 24 months
  This is an exploratory randomized sub-study with the objective of estimating the efficacy of CM24 and nivolumab with chemotherapy (Nal-IRI/5-FU/LV or gemcitabine/ nab-paclitaxel) and chemotherapy only (Nal- IRI/5-FU/LV or gemcitabine/nab-paclitaxel) as measured by overall survival.

SECONDARY OUTCOMES:
Maximum serum concentration [Cmax] | Up to 24 months
  Maximum serum concentration [Cmax] of CM24
Time of maximum concentration [Tmax] | Up to 24 months
  Time of maximum concentration [Tmax] of CM24
Area under the serum concentration curve [AUC] | Up to 24 months
  Area under the serum concentration curve [AUC] of CM24
Half life | Up to 24 months
  Half life of CM24
Drug clearance | Up to 24 months
  Drug clearance of CM24
Volume of distribution | Up to 24 months
  Volume of distribution of CM24
Serum ADA parameters | Up to 24 months
  Serum ADA parameters of CM24 as measured by percentage of patients who are positive for the presence of anti-drug antibodies
Objective Response Rate when CM24 is used in combination with nivolumab | Up to 24 months
Disease Control Rate when CM24 is used in combination with nivolumab | Up to 24 months
Median Duration of Response when CM24 is used in combination with nivolumab | Up to 24 months
Median Time to Response when CM24 is used in combination with nivolumab | Up to 24 months
Progression Free Survival when CM24 is used in combination with nivolumab | Up to 48 months
Overall Survival when CM24 is used in combination with nivolumab | Up to 48 months
Population pharmacokinetics when CM24 is used in combination with nivolumab as measured by the maximum plasma concentration [Cmax] | Up to 24 months
Population pharmacokinetics when CM24 is used in combination with nivolumab as measured by the average area under the concentration curve [AUC] | Up to 24 months
Population pharmacokinetics when CM24 is used in combination with nivolumab as measured by the median area under the concentration curve [AUC] | Up to 24 months
Population pharmacokinetics when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV as measured by the maximum plasma concentration [Cmax] | Up to 24 months
Population pharmacokinetics when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV as measured by the average area under the concentration curve [AUC] | Up to 24 months
Population pharmacokinetics when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV as measured by the median area under the concentration curve [AUC] | Up to 24 months
Disease Control Rate when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV | Up to 24 months
Duration of Response when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV | Up to 24 months
Time to Response when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV | Up to 24 months
Progression Free Survival when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV | Up to 48 months
Overall Survival when CM24 is used in combination with nivolumab and gemcitabin/nab-paclitaxel or Nal-IRI/5-FU/LV | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schickler, PhD, Study Director — Famewave Ltd.
Locations (18):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Sheba Medical Center, Ramat Gan
- Spain (11):
  - Hospital Clinic Barcelona, Barcelona
  - NEXT Oncology Barcelona, Barcelona
  - Vall d' Hebron Institute of Oncology (VHIO), Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital South Texas Accelerated Research Therapeutics (START) Madrid - CIOCC, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - NEXT Oncology Madrid, Pozuelo de Alarcón
  - Hospital Quiron Salud Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No